CLINICAL TRIAL: NCT04312815
Title: A Randomized,Placebo Controlled, Double-blind, Parallel Group, Phase III Study to Evaluate the Efficacy and Safety of SM03, Compared to Placebo, in Patients With Moderate-to-Severely Active Rheumatoid Arthritis Receiving Methotrexate
Brief Title: A Study Assessing the Efficacy and Safety of SM03 in Patients With Active Rheumatoid Arthritis Receiving MTX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM03-RA-III-V4.0
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis(RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SM03 600 mg (Experimental): SM03: 600 mg intravenous (IV) Randomizd period:on week 0,2,4 and 12,14,16;Participants with inadequate response (defined as less than 10% improvement from baseline in TJC and SJC by Week 12) were rescued with open label SM03 600 mg IV treatment.
  Open-lable treatment on week 24,30,36,42,48; Methotrexate: 7.5-20 mg/wk oral.
  Interventions: Drug: SM03; Drug: MTX
- Placebo (Placebo Comparator): placebo: 600 mg intravenous (IV) on week 0,2, 4, and week 12,14,16;Participants with inadequate response (defined as less than 10% improvement from baseline in TJC and SJC by Week 12) were rescued with open label SM03 600 mg IV treatment.
  SM03: 600 mg intravenous (IV) on week 24,30,36,42,48; Methotrexate: 7.5-20 mg/wk oral.
  Interventions: Drug: SM03; Drug: Placebo; Drug: MTX

INTERVENTIONS:
Drug: SM03 — SM03: 600 mg intravenous (IV)
Drug: Placebo — Placebo: 600 mg intravenous (IV)
  Arms: Placebo
Drug: MTX — Methotrexate: 7.5-20 mg/wk oral

SUMMARY:
* To demonstrate that SM03 added to methotrexate (MTX) reduce signs and symptoms of rheumatoid arthritis (RA) in Chinese RA participants with an inadequate response to MTX.
* To assess the safety of SM03 added to MTX in Chinese RA participants with an inadequate response to MTX

DETAILED DESCRIPTION:
The total duration of study was expected up to 58 weeks (screening period of 6 weeks, randomized treatment period of 24 weeks and open-label treatment extention period of 24 weeks , and a 4-week post treatment observation).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-75 years of age.
* Rheumatoid arthritis (RA) for ≥ 6 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria, or 2010 ACR/EULAR for the classification of rheumatoid arthritis.
* Moderate to severe active RA with swollen joint count (SJC) ≥ 6(66 joint count), and tender joint count (TJC) ≥ 8 (68 joint count) at screening and baseline.
* At screening, either High sensitivity C-Reactive Protein (hs-CRP) ≥ 1.5 UNL, or Erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour, or Morning stiffness of joint for ≥ 45 minutes.
* Inadequate response to methotrexate, having received and tolerated at a dose of 7.5-20 mg/week for ≥ 12 weeks, at a stable dose over the past 4 weeks.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA.
* Use of any biological DMARDs for RA.
* Concurrent treatment with any Disease Modifying Anti-Rheumatic Drug (DMARD) other than methotrexate
* Active infection, or history of serious or chronic infection

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24 | Week 24
  To achieve an ACR20 required at least a 20% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 20% improvement in three of the following five additional measurements:
  Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]); Patient's global assessment of disease activity (assessed using a 10 cm VAS); Patient's assessment of pain (assessed using a 10 cm VAS); Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3); Acute phase reactant: C-reactive protein (CRP)

SECONDARY OUTCOMES:
Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 12,52 | Week 12,52
  To achieve an ACR20 required at least a 20% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 20% improvement in three of the following five additional measurements:
  Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]); Patient's global assessment of disease activity (assessed using a 10 cm VAS); Patient's assessment of pain (assessed using a 10 cm VAS); Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3); Acute phase reactant: C-reactive protein (CRP)
Percentage of Participants With an ACR50/ACR70 Response at Week 12,24,52 | Week 12,24,52
  To achieve an ACR50/ACR70 required at least a 50%/70% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 50%/70% improvement in three of the following five additional measurements:
  Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]); Patient's global assessment of disease activity (assessed using a 10 cm VAS); Patient's assessment of pain (assessed using a 10 cm VAS); Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3); Acute phase reactant: C-reactive protein (CRP)
Change From Baseline in Disease Activity Score (DAS28-ESR) at Week 12,24,52 | Baseline and Week12,24,52
  The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  The number of swollen and tender joints assessed using the 28-joint count; Erythrocyte sedimentation rate (ESR); Patient's global assessment of disease activity measured on a 10 cm visual analog scale.
  The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 12,24,52 | Baseline and Week12,24,52
  A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity.
  A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score of less than or equal to 3.2.
  A Moderate Response is defined as either:
  an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 from Baseline and attainment of a DAS28 score of less than or equal to 5.1 or, an improvement (decrease) in the DAS28 of more than 1.2 from Baseline and attainment of a DAS28 score of greater than 3.2.
  No Response is defined as either an improvement (decrease) in the DAS28 of less than or equal to 0.6, or an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 of more than 5.1.
Percentage of Participants With Adverse Events | For Placebo arm: Baseline up to week 24; For SM03 arm: Baseline up to week 52;
  Percentage of participants who reported an AE or SAE, a drug-related AE, who had an acute infusion reaction, an AE leading to study drug discontinuation, with an infection or serious infection, or who died.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, MD, Principal Investigator — Department of Rheumatology and Immunology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hostipal, Beijing, China

REFERENCES:
- [Derived] Wong KL, Li Z, Ma F, Wang D, Song N, Chong CH, Luk KK, Leung SO. SM03, an Anti-CD22 Antibody, Converts Cis-to-Trans Ligand Binding of CD22 against alpha2,6-Linked Sialic Acid Glycans and Immunomodulates Systemic Autoimmune Diseases. J Immunol. 2022 Jun 15;208(12):2726-2737. doi: 10.4049/jimmunol.2100820. Epub 2022 Jun 10. PMID 35688465